CLINICAL TRIAL: NCT04886427
Title: Implementation of a Multidimensional Quality Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Sint-Trudo Hospital (Other)
Responsible Party: Principal Investigator, Kris Vanhaecht, Professor, KU Leuven
Other Study IDs: IMQM
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Management Systems; Quality Improvement; Public Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quickscan for patients and their kin: Patients and/or kin who are treated in the hospitals will be invited to fill in the quickscan.
  Interventions: Other: No intervention
- Quickscan for healthcare professionals: Healthcare professionals working in the hospitals will be invited to fill in the quickscan.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Measure the experiences of the current care

SUMMARY:
The aim of this study is to measure the experiences about the current care of the patients, their kin and staff by a quickscan based on a multidimensional quality model. Further more we want to define the psychometric characteristics of the quickscan.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Treated/working in the hospital

Exclusion Criteria:

* Do not understand Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Treated or working in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Perception of the organisation of care | During their treatment or work experience in the hospital
  Patients, kin and healthcare professionals will give their perception regarding the organisation of care

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - UZ Leuven, Leuven
  - Sint-Trudo Ziekenhuis, Sint-Truiden
  - RZ Heilig Hart, Tienen

IPD SHARING:
Plan to Share IPD: No